CLINICAL TRIAL: NCT04066413
Title: Growth and Tolerance Trial in Healthy Infants on Infant Formula Supplemented With a Human Milk Oligosaccharide
Brief Title: Growth and Tolerance Trial on Infant Formula With HMO
Acronym: Stardust
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recruitment difficulties
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stardust
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy Growth
Keywords: infant formula; human milk oligosaccharide; HMO; growth
MeSH Terms: interventions — Health Maintenance Organizations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breastfed group (No Intervention): Non-randomized breastfed reference group
- Control formula (Placebo Comparator): Group receiving standard infant formula
  Interventions: Other: Standard infant formula
- Formula with HMO (Active Comparator): Group receiving standard infant formula supplemented with HMO
  Interventions: Other: Infant formula supplemented with HMO

INTERVENTIONS:
Other: Standard infant formula — Standard infant formula
  Arms: Control formula
Other: Infant formula supplemented with HMO — Infant formula supplemented with HMO
  Arms: Formula with HMO

SUMMARY:
The aim of the study is to compare growth of healthy infants fed an infant formula supplemented with a human milk oligosaccharide to that of infants on standard formula.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 37 weeks
* Birth weight ≥ 2500 grams
* No recognized diseases (such as cardiac, pulmonary, gastrointestinal, renal or genetic diseases)
* Boys and girls
* Recruited < 1 month/age
* Being available for follow up until the age of 4 months
* Exclusive formula feeding or exclusive breast feeding at time of recruitment

Exclusion Criteria:

* Gestational age <37 weeks
* Birth weight <2500 grams
* Severe acquired or congenital diseases, mental or physical disorders
* Illness at screening/ inclusion
* Incapability of parents/caregivers to comply with the study protocol
* Received antibiotics within the first month of life
* Not tolerating standard cow's milk based infant formula
* Participation in another clinical trial
* Maternal illicit drug use during pregnancy or post-partum period
* Parent/caregiver does not have a cell phone to use for filling out questionnaires

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 265 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Growth | From enrollment until end of the 3 month-study
  Infant growth measured as body weight gain per day

SECONDARY OUTCOMES:
Weight | Monthly, from enrollment until end of the 3 month-study
  Infant weight (kg)
Recumbent length | Monthly, from enrollment until end of the 3 month-study
  Infant length (cm and cm/day)
Head circumference | Monthly, from enrollment until end of the 3 month-study
  Head circumference (cm and cm/day)
Anthropometry z-scores | Monthly, from enrollment until end of the 3 month-study
  World Health Organization (WHO) growth standard calculated z-scores for weight, length, weight-for-length and head circumference
Formula tolerance | Monthly, from enrollment until end of the 3 month-study
  Parents are asked to keep a diary on formula intake 3 days prior to each monthly study visit
Gastro-intestinal comfort | Monthly, from enrollment until end of the 3 month-study
  Parents are asked to keep a diary 3 days prior to each monthly study visit including questions on gastro-intestinal symptoms (e.g. cramps, constipation, vomiting) and crying behavior

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No